CLINICAL TRIAL: NCT04800185
Title: Characterizing Skin Microbiome Change in Atopic Dermatitis Patients After Targeted Topical Treatment Using Crisaborole Ointment
Brief Title: Characterizing Skin Microbiome Change in Atopic Dermatitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Natasha Mesinkovska, Prinicipal Investigator, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20195479
Record Dates: First submitted 2021-03-05; First posted 2021-03-16 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema
Keywords: skin microbiome; crisaborole
MeSH Terms: conditions — Dermatitis, Atopic | interventions — crisaborole

STUDY DESIGN:
Intervention Model Description: Subjects will function as their own internal control with one lesion left untreated
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment group (Other)
  Interventions: Drug: Crisaborole 2% Top Oint; Genetic: Skin Microbiome Swabs

INTERVENTIONS:
Drug: Crisaborole 2% Top Oint — To analyze the skin microbiome of patients with atopic dermatitis before, during, and after treatment with crisaborole 2% ointment
Genetic: Skin Microbiome Swabs — At the baseline visit the investigator will identify sites for swabbing the skin including one affected distinct crisaborole-treated AD lesion, and one untreated AD lesion. The lesions will both be sampled at baseline, 14 days into treatment, 28 days into treatment, 3 months into treatment, and 4 weeks after treatment completion. Photographs of each lesion will be taken for reference. Skin swabs will be obtained in a sterile fashion using a BD Culture SwabsTM EZ Collection and Transport System (or equivalent) and soaked with sterilized 0.15 M NaCl and 0.1% Tween-20. The samples will be frozen at -80 C, kept at this temperature, and stored until analysis may be completed.

SUMMARY:
Atopic dermatitis (AD), also known as eczema, is an inflammatory disease of the skin affecting a large proportion of the pediatric and adult patient population. Chronic itching and eczematous lesions lead to a high burden of disease and associated patient morbidity with higher infection rates, emotional stress and associated psychological disease. The microbiome community contributes to human health through several mechanisms. Current research suggests that derangements in the normal microbiota may lead to inflammatory bowel disease, allergy, and metabolic syndromes. Specific to dermatology, new literature has demonstrated that changes in the microbiome may play a role in the development of atopic dermatitis.

With this study, the investigators hope to characterize the baseline atopic dermatitis skin microbiome and monitor the evolution of the participants skin microbiome during and after treatment with anti-inflammatory topical medications, specifically the Food and Drug Administration (FDA)-approved phosphodiesterase inhibitor, crisaborole ointment 2% (Eucrisa).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 2 years or older at the time of consent.
2. Patients may be male or female.
3. Patients may have any skin phototype.
4. Patients with a clinical diagnosis of atopic dermatitis according to the Hanifin and Rajka criteria. Atopic dermatitis diagnosis must be stable at least for 1 month per caregiver or patient.
5. Atopic dermatitis affecting at least 5% of the patient's body surface area with at least two distinct lesional sites.
6. Atopic dermatitis must meet a score of mild to moderate on the baseline Investigator's Static Global Assessment (iSGA).
7. If greater than or equal to 18 years old at the time of consent, is able to provide written informed consent and will comply with all study procedures. If less than 18 years old at the time of consent, parent or guardian is able to provide written informed consent with all children greater than or equal to 7 years old at the time of consent also providing written assent, and will comply with all study procedures.

Exclusion Criteria:

1. Patients less than 2 years old at the time of consent.
2. Patients unable to provide written informed consent.
3. Patients must not have used systemic biologic therapy, systemic immunosuppressive therapy, or systemic immunomodulating therapy within three months of baseline visit.
4. Patients must not have had phototherapy within three months of baseline visit.
5. Patients must not have used topical corticosteroids or topical calcineurin inhibitor within 28 days of baseline visit.
6. Patients must not have previously been treated with topical phosphodiesterase-4 inhibitor.
7. Patients must not have a known hypersensitivity reaction to crisaborole or any of its known vehicle components.
8. Patients must not have any active skin infection at the time of screening.
9. Patients must not have any other overlying inflammatory disease such as psoriasis.
10. Patients must not be currently pregnant, breastfeeding or planning pregnancy during the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
To determine a change in skin microbiome taxonomic units after 16 weeks of treatment with Crisaborole in atopic dermatitis. | 16 weeks
  To analyze the atopic dermatitis microbiome using advanced genomic techniques after treatment with topical PDE4 inhibitors. Using 16S library preparation, sequencing, merging of MiSeq paired-end sequence reads, and identification of operational taxonomic units, the investigators hope to identify the bacterial and fungal content of skin microbiome samples from 20 AD participants before and after treatment with crisaborole at a total of 6 visits over 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Atanaskova Mesinkovska, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine - Dermatology Clinical Research, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No